CLINICAL TRIAL: NCT03772431
Title: A Randomized Controlled Trial of Narrative Voice and Introduction Content to Improve Interactive Voice Response (IVR) Survey Performance in Bangladesh and Uganda
Brief Title: Use of Narrative Voice and Introduction Content to Improve Interactive Voice Response Surveys in Bangladesh and Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: The Bloomberg Family Foundation, Inc. (Other); Makerere University (Other); Institute of Epidemiology, Disease Control and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318-3
Record Dates: First submitted 2018-12-10; First posted 2018-12-11 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2018-12

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; narration
MeSH Terms: conditions — Noncommunicable Diseases; Narration

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of four narrator/introduction combinations: 1) male voice, informational content; 2) male voice, motivational content; 3) female voice, informational content; 4) female voice, motivational content.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Male Informational (Experimental): Male voice, informational introduction
  Interventions: Other: Male Voice; Other: Informational Introduction
- Male Motivational (Experimental): Male voice, motivational introduction
  Interventions: Other: Motivational Introduction; Other: Male Voice
- Female Informational (Experimental): Female voice, informational introduction
  Interventions: Other: Female Voice; Other: Informational Introduction
- Female Motivational (Experimental): Female voice, motivational introduction
  Interventions: Other: Female Voice; Other: Motivational Introduction

INTERVENTIONS:
Other: Female Voice — The survey was narrated by a female voice
  Arms: Female Informational; Female Motivational
Other: Motivational Introduction — The survey introduction was worded to include motivational content
  Arms: Female Motivational; Male Motivational
Other: Male Voice — The survey was narrated by a male voice
  Arms: Male Informational; Male Motivational
Other: Informational Introduction — The survey introduction was worded to include informational content
  Arms: Female Informational; Male Informational

SUMMARY:
This study evaluates the effect of two different narrative voices (one male and one female) and two different introductions (one with informational content and the other with additional motivational content) on interactive voice response (IVR) survey cooperation, response, refusal, and contact rates, as compared to a control group (male, informational), in Bangladesh and Uganda.

DETAILED DESCRIPTION:
Using random digit dialing (RDD) sampling techniques, participants were randomized to one of four arms: 1) male narrator and informational survey introduction, 2) male narrator and motivational survey introduction, 3) female narrator and informational survey introduction, and 4) female narrator and motivational survey introduction,male motivational, female informational, female motivational) which were then followed by a noncommunicable disease risk factor survey. This mobile phone survey was sent as an interactive voice response (IVR). In IVR surveys, participants use their touch tone key pad to answer pre-recorded questions. (i.e. If you are male, press 1; if you are female, press 2). This study was conducted in both Bangladesh and Uganda.

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Bangladesh, conversant in either English or Bangla language. In Uganda, conversant in either Luo, Luganda, Runyakitara or English languages.

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5580 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2017-07-17 (Actual); Study Completion 2017-07-17 (Actual)

PRIMARY OUTCOMES:
Cooperation rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, cooperation rate is defined as I/(I+P+R) where I is complete interviews, P is partial interviews, and R is refusals and breakoffs
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, response rate is defined as (I+P)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns.

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, refusal rate is defined as (R)/(I+P+R+eU) where R is refusals and breakoffs, I is complete interviews, P is partial interviews, and eU is the estimated eligible proportion of unknowns
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research, contact rate is defined as (I+P+R)/(I+P+R+eU) where I is complete interviews, P is partial interviews, R is refusals and breakoffs, and eU is the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, PhD, MBBS, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health; George W. Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Institute of Epidemiology Disease Control and Research, Dhaka, Bangladesh
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722
- [Derived] Labrique A, Nagarajan M, Kibria GMA, Vecino-Ortiz A, Pariyo GW, Ali J, Kaufman MR, Gibson D. Improving success of non-communicable diseases mobile phone surveys: Results of two randomized trials testing interviewer gender and message valence in Bangladesh and Uganda. PLoS One. 2023 May 24;18(5):e0285155. doi: 10.1371/journal.pone.0285155. eCollection 2023. PMID 37224125